CLINICAL TRIAL: NCT07071948
Title: A Single-Center Clinical Study on the Efficacy and Safety of Vortex Intelligence Stone Optimized Removal (VISOR)
Brief Title: A Single-Center Clinical Study on the Efficacy and Safety of VISOR
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2025-0324
Record Dates: First submitted 2025-07-14; First posted 2025-07-18 (Actual); Last update posted 2025-09-26 (Actual); Status verified 2025-07

CONDITIONS: Urolithiasis, Calcium Oxalate; Kidney Stone
Keywords: urolithiasis; kidney stone; stone free rate; VISOR
MeSH Terms: conditions — Nephrolithiasis, Calcium Oxalate; Kidney Calculi; Urolithiasis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- VISOR Treatment (Experimental): All enrolled participants (n=20) will undergo upper urinary tract stone removal using the investigational device VISOR (Vortex Intelligence Stone Optimized Removal). The procedure includes:
  1. Integrated irrigation-aspiration and real-time pressure monitoring/control (safety threshold: <30 mmHg).
  2. Holmium laser lithotripsy with simultaneous stone fragment removal.
  3. Postoperative assessment:
  Urinary CT scan at 24h to determine immediate stone-free rate (residual stones <4 mm).
  Follow-up imaging (CT/ultrasound) and complication monitoring at 28±7 days.
  Interventions: Device: Multifunctional Integrated Flexible Ureteroscope

INTERVENTIONS:
Device: Multifunctional Integrated Flexible Ureteroscope — Investigational ureteroscope with three integrated functions:
  1. Real-time pressure control: Continuous renal pelvic pressure monitoring with auto-adjustment of irrigation/aspiration flow to maintain pressure <30 mmHg (safety threshold)
  2. Simultaneous lithotripsy & fragment removal: Holmium laser lithotripsy (200-365 μm fiber) coordinated with suction through working channel
  3. Single-pass stone clearance: Designed to reduce residual fragments requiring secondary procedures
  Distinguishing features vs conventional ureteroscopes:
  1. Eliminates need for separate suction devices
  2. Prevents intraoperative "washout failure" causing obscured vision
  3. Patent-pending pressure sensor
  Other Names: Xinwell Scope

SUMMARY:
Goal of this trial:

To test a new tool called VISOR in adults (aged 18-80) with 1-3 cm kidney or ureter stones. We want to see:

1. If it's safe and works well
2. If its built-in features (flushing/suction, pressure control, and stone-breaking/removal) help clear stones better while keeping surgery safe.

Main questions:

1. Can the VISOR clear stones successfully (with fragments <4 mm left) for at least 9 out of every 10 people within 24 hours after surgery?
2. Will serious problems (like severe infections or ureteral injuries) happen to no more than 1 in 20 people (5%)?
3. Can the device keep pressure inside the kidney below 30 mmHg (a safe level) during the entire surgery?

What participants will do:

Have stone removal surgery using VISOR (breaks and removes stones at the same time).

Get a CT scan within 24 hours after surgery to check if stones are cleared.

Return 4 weeks (±1 week) after surgery for:

An imaging test (CT or ultrasound)

A check for any health problems related to the surgery.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with upper urinary tract calculi, where the maximum diameter of a single calculus or the cumulative diameter of multiple calculi is 1-3 cm
2. Patients who choose to undergo "flexible ureteroscopic holmium laser lithotripsy"
3. Aged 18-80 years, regardless of gender
4. Subjects without mental illness or language dysfunction, who can understand the details of this study and sign the informed consent form

Exclusion Criteria:

1. Patients with ureteral stricture or a history of ureteral stricture
2. Patients with a history of open renal and/or ureteral surgery or laparoscopic surgery
3. Fever (body temperature ≥ 38℃) due to urinary tract infection or other reasons within one week before surgery
4. Pregnant women, lactating women, or women who are in the menstrual period
5. ASA classification > Grade 3: patients with severe systemic diseases, heart diseases, pulmonary insufficiency, and failure of important organ functions, etc., who cannot tolerate anesthesia or surgery
6. Patients with anatomical malformations such as polycystic kidney, horseshoe kidney, and ectopic kidney
7. Patients with abnormal coagulation function (e.g., international normalized ratio (INR) > 1.5 or platelet count < 80 × 10⁹/L)
8. Patients with failed sheath placement during surgery

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-08-06 (Actual); Primary Completion 2025-10-31 (Estimated); Study Completion 2027-02-28 (Estimated)

PRIMARY OUTCOMES:
24-hour stone-free rate after Xinwell Scope lithotripsy | within 24 hours postoperatively
  Proportion of participants with complete stone clearance (defined as no residual fragment ≥4 mm in maximum diameter) assessed by non-contrast urinary CT scan within 24 hours post-surgery. Calculated as:
  (Number of patients with residual stones <4 mm / Total analyzed participants) × 100% Significance: Directly evaluates the device's integrated suction function for real-time fragment removal during the procedure.

SECONDARY OUTCOMES:
1-month stone-free rate | 28±7 days postoperatively
  Proportion of participants with residual stones <4 mm assessed by CT (if baseline residual ≥4 mm) or renal ultrasound (if no baseline residual) at 28±7 days post-surgery.
Operative time | During surgery
  Duration (minutes) from initial ureteroscope insertion to final removal.
Intraoperative renal pelvic pressure | Continuous monitoring during lithotripsy
  Mean/Max pressure (mmHg) recorded by built-in sensor. Safety target: <30 mmHg.
Ureteral injury rate | During surgery
  Graded via intraoperative video review:
  Grade 0: Mucosal bleeding only
  Grade 1-4: Mucosal to full-thickness injury
Postoperative complication rate | 24h, 28 ±7 days , 1 month
  Includes:
  Fever (>38.0°C within 24h)
  Clavien-Dindo grade ≥II complications
  Ureteral stenosis (imaging-confirmed at 1 months)

CONTACTS AND LOCATIONS:
Overall Officials: Bohan Wang, MD., Ph.D, Principal Investigator — 2nd Affiliated Hospital, School of Medicine, Zhejiang University, China
Locations (1):
- 2nd Affiliated Hospital, School of Medicine, Zhejiang University, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No
1. Intellectual Property Protection
     * The investigational device (Xinwell Scope) contains patent-pending technologies owned by Ningbo Xinwell Medical Technology Co., Ltd.
     * Public disclosure of raw performance data (e.g., real-time pelvic pressure metrics) may compromise proprietary algorithms.
  2. Privacy Risks of De-identified Data
     * Key datasets (intraoperative videos, dynamic pressure recordings) carry re-identification risks despite de-identification.